CLINICAL TRIAL: NCT01934335
Title: A Randomized, Double-Blind, Placebo-Controlled Trial Investigating the Effect of Vandetanib on Cellular Markers of Proliferation and Apoptosis in Invasive Breast Cancer
Brief Title: Effect of Vandetanib on Cellular Markers in Invasive Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drugs unavailable
Sponsor: Ronald Weigel (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Ronald Weigel, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201301763
Record Dates: First submitted 2013-08-29; First posted 2013-09-04 (Estimated); Results first posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Invasive Breast Cancer
Keywords: breast cancer, TKI, tyrosine kinase inhibitor, vandetanib, Ki-67
MeSH Terms: conditions — Breast Neoplasms | interventions — vandetanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vandetanib (Experimental): Vandetanib, 300 mg, PO, q day for 7-14 days prior to surgery
  Interventions: Drug: Vandetanib
- Placebo (Placebo Comparator): Placebo, PO, q day for 7-14 days prior to surgery.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vandetanib
  Other Names: ZD6474
  Arms: Vandetanib
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this project is to examine whether treatment with vandetanib has an effect on the tumor cells in breast cancer by examining tissue markers.

DETAILED DESCRIPTION:
The purpose of this research study is to test whether vandetanib has an effect on tumor growth markers. Vandetanib is not approved by the FDA for use in treating breast cancer. This study will compare vandetanib to a placebo.

The proposed study is designed to determine the change in Ki-67 expression on paired breast cancer samples obtained before and after treatment with vandetanib. Other tumor markers including RET, TUNEL and phosphorylation specific levels of ERK1/2, AKT and mTOR will also be assessed on the paired samples.

Those who have a core biopsy of the breast which demonstrates invasive breast cancer and requires surgical excision of the lesion will be eligible for inclusion in the study. The tyrosine kinase inhibitor, vandetanib 300 mg, will be given once a day for 7-14 days prior to surgery. Following surgery, tissue markers would be analyzed on each of the paired samples, allowing for rapid assessment of in vivo response to TKI treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with core breast biopsy that, on pathology review, demonstrates invasive breast cancer and are determined to need surgical excision of the lesion. All subtypes of invasive breast cancer will be enrolled. Core biopsy specimens of enrolled patients will be stained for RET by immunohistochemistry and scored, however, patients will not be excluded according to RET expression.
* Female gender
* Age >/= 18 years of age
* ECOG performance status </= 2
* Life expectancy of greater than 6 months
* Ability and willingness to provide informed consent to participate in study

Exclusion Criteria:

* Prolonged QT interval (QTc > 480 milliseconds) on screening EKG or congenital long QT syndrome
* Any concomitant medications that are known to be associated with Torsades de Pointes or QT elongation (see appendix 2).
* Hypertension not controlled by medical therapy (systolic BP greater than 160 millimeters of mercury [mmHg] or diastolic blood pressure great than 100 mmHg).
* Patients taking metformin or digoxin.
* History of arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia), which is symptomatic or requires treatment (CTCAE Grade 3), symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia. Patients with atrial fibrillation controlled by medication are permitted.
* Significant cardiac event (e.g., myocardial infarction), superior vena cava syndrome, New York Heart Association (NYHA) classification of heart disease ≥2 within 12 weeks, or presence of cardiac disease that in the opinion of the Investigator increases the risk of ventricular arrhythmia.
* Serum calcium or magnesium outside the institutional range of normal.
* Serum Potassium < 4.0 mmol/L or above 5.0 mmol/L
* Creatinine clearance < 50 ml/min
* PT > 12 seconds or PTT > 31 seconds
* Platelet count of < 100,000
* Serum bilirubin greater than 1.5 mg/dl
* Alanine aminotransferase (ALT) > 50 U/L, aspartate aminotransferase (AST) > 65 U/L, or alkaline phosphatase (ALP) > 250 U/L
* Any cytotoxic treatments, such as neoadjuvant chemotherapy, planned before subsequent surgical procedure.
* Previous exposure to Vandetanib
* Previous enrollment or randomization in this study
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and staff at UIHC).
* Previous or current malignancies of other histologies within the last 5 years, with the exception of in situ carcinoma of the cervix, and adequately treated basal cell or squamous cell carcinoma of the skin.
* Patients who have received prior surgical site radiation.
* Patients on CYP3A4 inhibitors or inducers (see appendix 1).
* Inability to test core biopsy for study markers
* Pregnancy or lactation at the time of study entry. (Note: Pregnancy testing must be performed within 2 weeks prior to randomization according to institutional standards for women of childbearing potential.)

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronal Weigel, MD, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Vandetanib: Vandetanib, 300 mg, PO, q day for 7-14 days prior to surgery
  Vandetanib
- Placebo: Placebo, PO, q day for 7-14 days prior to surgery.
  Placebo
Period: Overall Study
Arm/Group | Vandetanib | Placebo
Started | 7 | 5
Completed | 6 | 4
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Subjects who have a core biopsy of the breast which demonstrates invasive breast cancer and require surgical excision of the lesion are eligible for inclusion in the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Vandetanib | Placebo | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Full Range); unit: years] | 55.5 [35.5 to 71.1] | 62.9 [45.4 to 72.5] | 58.8 [35.5 to 72.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 5 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 5 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Ki-67 Cells Observed 2 Weeks Post-treatment
Description: Pre- and post-treatment samples will be assessed by immunohistochemistry for positivity for Ki-67.
Time Frame: 2 weeks
Population: 10 subjects took study drug and completed surgery
Measure: Mean (Standard Deviation); unit: percentage of positivity for Ki-67.
Arm/Group | Vandetanib | Placebo
Number analyzed (Participants) | 6 | 4
percentage of positivity for Ki-67. | 0.3 (0.08) | 2 (0.05)
Statistical Analysis 1: Comparison: Vandetanib vs Placebo; Test type: Superiority; p = 0.51, t-test, 2 sided

2. Secondary Outcome: Percent Change From Baseline in TUNEL Observed 2 Weeks Post-treatment
Description: Pre- and post-treatment samples will be assessed by immunohistochemistry for positivity for TUNEL.
Time Frame: 2 weeks
Population: 10 subjects took study drug and completed surgery
Measure: Mean (Standard Deviation); unit: percentage of for positivity for TUNEL
Arm/Group | Vandetanib | Placebo
Number analyzed (Participants) | 6 | 4
percentage of for positivity for TUNEL | 0.48 (0.71) | 1.02 (89)
Statistical Analysis 1: Comparison: Vandetanib vs Placebo; Test type: Superiority; p = 0.35, t-test, 2 sided

3. Other Pre Specified Outcome: Percent Change From Baseline in RET Expression Observed 2 Weeks Post-treatment
Description: Results will be stratified by RET gene expression, a negative prognostic indicator in breast cancer, to demonstrate that RET is a marker of response.
Time Frame: 2 weeks
Population: 6 patients that got the study drug and completed surgery by RET expression were analyzed
Measure: Mean (Standard Deviation); unit: percent change of RET positive samples
Arm/Group | Vandetanib | Placebo
Number analyzed (Participants) | 3 | 3
percent change of RET positive samples
  Ki-67 | -0.3 (0.03) | 1.0 (0.12)
  TUNEL | 0.77 (0.32) | 0.2 (0.12)
Statistical Analysis 1: Comparison: Vandetanib vs Placebo; Test type: Superiority; p = 0.43, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Vandetanib | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 5/6 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vandetanib (N=6) | Placebo (N=5)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Dehydration (General disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Hot flashes (General disorders) | 1 (1) | 0 (0)
Dysgeusia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Itchy eyes (Eye disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-05): https://cdn.clinicaltrials.gov/large-docs/35/NCT01934335/Prot_SAP_000.pdf
  • Informed Consent Form (2018-09-04): https://cdn.clinicaltrials.gov/large-docs/35/NCT01934335/ICF_001.pdf